CLINICAL TRIAL: NCT03811301
Title: Neurodevice Phase I: Wireless Implantable Neurodevice Microsystem for Neuroprosthesis and Neuroscience
Brief Title: [BrainConnexion] - Neurodevice Phase I Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Neuroscience Institute (Other)
Collaborators: Institute of Microelectronics (Unknown); Institute of Molecular and Cell Biology (Unknown); Institute for Infocomm Research (Other); Nanyang Technological University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BrainConnexion
Record Dates: First submitted 2018-12-17; First posted 2019-01-22 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2022-11

CONDITIONS: Tetraplegia; Tetraplegia/Tetraparesis; Spinal Cord Injuries; Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Locked-in Syndrome; Muscular Dystrophies
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries; Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Locked-In Syndrome; Muscular Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Interventional (Experimental): Wireless Implantable Neurodevice Microsystem
  Interventions: Device: BrainConnexion

INTERVENTIONS:
Device: BrainConnexion — A 4.4mm by 4.2mm electrode array is placed onto the surface of the motor cortex which is then connected to a miniaturized neural recording microsystem that transmits signals wirelessly to control an external assistive device. Neural signals are recorded at least once every week for 12 months or longer.
  Other Names: Neurodevice; NeuroPort

SUMMARY:
This study aims to evaluate the safety of a wireless implantable neurodevice microsystem in tetraplegic patients, as well as the efficacy of the electrodes for long-term recording of neural activities and the successful control of an external device.

DETAILED DESCRIPTION:
The goal of this study is to develop a miniaturized wireless implantable neurodevice microsystem that records and transmits signals from the motor cortex of tetraplegic patients, bypassing the damaged nervous tissue, to control an external assistive device that restores some form of independence to patients in terms of communication or mobility.

ELIGIBILITY:
Inclusion Criteria:

1. 21 years old and older
2. Tetraparesis
3. Written informed consent obtained from the patient or legal representative (in the event where the patient is unable to provide consent) prior to entry into the study in accordance with local EC/IRB regulations and/or other application regulations for surrogate consent.
4. Able to perform the pre-operation Brain Computer Interface training as judged by the research team.

Exclusion Criteria:

1. Significant medical co-morbidities e.g. cardiac disease
2. Bleeding disorders
3. Any contraindication to surgery
4. Other concomitant intracranial pathologies
5. History of seizures or epilepsy disorder
6. Complications of coagulopathy
7. Surgically unfit
8. Significant psychological issues e.g. Depression
9. Poor psychological support
10. Pregnancy
11. No means of communication
12. Any disease, in the opinion of the Investigator, that is unstable or which could jeopardise the safety of the patient

If applicable, psychological assessment may be performed prior to selection as the implantation process will be a long a stressful event, requiring a significant degree of patient cooperation and resilience.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-08-27 (Estimated)

PRIMARY OUTCOMES:
The number of serious adverse events (SAEs) and adverse events (AEs) reported per patient 12 months post-implantation. | 6 months post-implant
  The primary objective of this study is to determine the safety of the device. This will be assessed based on the number of SAEs and AEs reported for each patient during the 12 months post-implantation evaluation. This measure will considered a success if the device is not removed for safety reasons within 12-months after implantation.

SECONDARY OUTCOMES:
The signal quality of the electrodes for long-term recording of neural signals. | Day 1 to Day 365 post-implant
  Signal quality will be measured by the number of channels with identifiable single units tracked across each day for 12 months.
Decoding accuracy per training session. | Day 1 to Day 365 post-implant
  Decoding accuracy will be measured in percentage (%).
Number of successful trials per session | Day 1 to Day 365 post-implant
  The number of successful trials per training session will be measured in percentage (%).
Time taken to complete each trial per session | Day 1 to Day 365 post-implant
  This will be measured in seconds (s).

CONTACTS AND LOCATIONS:
Locations (1):
- National Neuroscience Institute, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Libedinsky C, So R, Xu Z, Kyar TK, Ho D, Lim C, Chan L, Chua Y, Yao L, Cheong JH, Lee JH, Vishal KV, Guo Y, Chen ZN, Lim LK, Li P, Liu L, Zou X, Ang KK, Gao Y, Ng WH, Han BS, Chng K, Guan C, Je M, Yen SC. Independent Mobility Achieved through a Wireless Brain-Machine Interface. PLoS One. 2016 Nov 1;11(11):e0165773. doi: 10.1371/journal.pone.0165773. eCollection 2016. PMID 27802344
- [Background] Hochberg LR, Serruya MD, Friehs GM, Mukand JA, Saleh M, Caplan AH, Branner A, Chen D, Penn RD, Donoghue JP. Neuronal ensemble control of prosthetic devices by a human with tetraplegia. Nature. 2006 Jul 13;442(7099):164-71. doi: 10.1038/nature04970. PMID 16838014
- [Background] Hochberg LR, Bacher D, Jarosiewicz B, Masse NY, Simeral JD, Vogel J, Haddadin S, Liu J, Cash SS, van der Smagt P, Donoghue JP. Reach and grasp by people with tetraplegia using a neurally controlled robotic arm. Nature. 2012 May 16;485(7398):372-5. doi: 10.1038/nature11076. PMID 22596161
- [Background] Collinger JL, Wodlinger B, Downey JE, Wang W, Tyler-Kabara EC, Weber DJ, McMorland AJ, Velliste M, Boninger ML, Schwartz AB. High-performance neuroprosthetic control by an individual with tetraplegia. Lancet. 2013 Feb 16;381(9866):557-64. doi: 10.1016/S0140-6736(12)61816-9. Epub 2012 Dec 17. PMID 23253623
- [Background] Aflalo T, Kellis S, Klaes C, Lee B, Shi Y, Pejsa K, Shanfield K, Hayes-Jackson S, Aisen M, Heck C, Liu C, Andersen RA. Neurophysiology. Decoding motor imagery from the posterior parietal cortex of a tetraplegic human. Science. 2015 May 22;348(6237):906-10. doi: 10.1126/science.aaa5417. PMID 25999506
- [Background] Schwarz DA, Lebedev MA, Hanson TL, Dimitrov DF, Lehew G, Meloy J, Rajangam S, Subramanian V, Ifft PJ, Li Z, Ramakrishnan A, Tate A, Zhuang KZ, Nicolelis MA. Chronic, wireless recordings of large-scale brain activity in freely moving rhesus monkeys. Nat Methods. 2014 Jun;11(6):670-6. doi: 10.1038/nmeth.2936. Epub 2014 Apr 28. PMID 24776634
- [Background] Yin M, Borton DA, Komar J, Agha N, Lu Y, Li H, Laurens J, Lang Y, Li Q, Bull C, Larson L, Rosler D, Bezard E, Courtine G, Nurmikko AV. Wireless neurosensor for full-spectrum electrophysiology recordings during free behavior. Neuron. 2014 Dec 17;84(6):1170-82. doi: 10.1016/j.neuron.2014.11.010. Epub 2014 Dec 4. PMID 25482026
- [Background] Zaaroor M, Kosa G, Peri-Eran A, Maharil I, Shoham M, Goldsher D. Morphological study of the spinal canal content for subarachnoid endoscopy. Minim Invasive Neurosurg. 2006 Aug;49(4):220-6. doi: 10.1055/s-2006-948000. PMID 17041833
- [Background] Lee, K., Singh, A., He, J., Massia, S., Kim, B., & Raupp, G. (2004). Polyimide based neural implants with stiffness improvement. Sensors Actuators B Chem,102(1), 67-72. doi: 10.1016/j.snb.2003.10.018.
- [Background] Cheng, M. Y., Je, M., Tan, K. L., et al. (2013). A low-profile three-dimensional neural probe array using a silicon lead transfer structure. J Micromechanics Microengineering, 23(9), 095013. doi:10.1088/0960-1317/23/9/095013.
- [Background] Cheng, M. Y., Yao, L., Tan, K. L., Lim, R., Li, P., & Chen, W. (2014). 3D probe array integrated with a front-end 100-channel neural recording ASIC. J Micromechanics Microengineering, 24(12), 125010. doi:10.1088/0960-1317/24/12/125010.
- [Background] Zou, X., Liu, L., Cheong, J. H., et al. (2013). A 100-Channel 1-mW implantable neural recording IC. IEEE Trans Circuits Syst I Regul Pap, 60(10), 2584-2596. doi:10.1109/TCSI.2013.2249175.
- [Background] Christopher and Dana Reeve Foundation. Christopher and Dana Reeve Foundation. https://www.christopherreeve.org/. Published 2016.
- [Background] Technical specifications for short range devices - Issue 1 Rev 7, Apr 2013. https://www.ida.gov.sg/~/media/Files/PCDG/Licensees/StandardsQoS/RadiocomEquipStd/TSSRD.pdf
- [Background] Liu X, Zhou J, Wang C, et al. An Ultralow-Voltage Sensor Node Processor With Diverse Hardware Acceleration and Cognitive Sampling for Intelligent Sensing. IEEE Trans Circuits Syst II Express Briefs. 2015;62(12):1149-1153. doi:10.1109/TCSII.2015.2468927.
- [Background] Rebsamen B, Guan C, Zhang H, Wang C, Teo C, Ang MH Jr, Burdet E. A brain controlled wheelchair to navigate in familiar environments. IEEE Trans Neural Syst Rehabil Eng. 2010 Dec;18(6):590-8. doi: 10.1109/TNSRE.2010.2049862. Epub 2010 May 10. PMID 20460212
- [Background] Rosa So, Libedinsky C, Kai Keng Ang, Wee Chiek Clement Lim, Kyaw Kyar Toe, Cuntai Guan. Adaptive decoding using local field potentials in a brain-machine interface. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:5721-5724. doi: 10.1109/EMBC.2016.7592026. PMID 28269554
- [Background] So RQ, Xu Z, Libedinsky C., Ang KK, Toe KK, Yen SC, Guan CT (2015) Neural Representations of Movement during Brain-Controlled Self-Motion. Conf Proc 7th International IEEE EMBS Conference on Neural Engineering.
- [Background] Xu Z, Guan CT, So RQ, Ang KK, Toe KK. (2015) Motor Cortical Adaptation Induced by Closed-Loop BCI. Conf Proc 7th International IEEE EMBS Conference on Neural Engineering.
- [Background] Xu Z, So RQ, Toe KK, Ang KK, Guan C. On the asynchronously continuous control of mobile robot movement by motor cortical spiking activity. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:3049-52. doi: 10.1109/EMBC.2014.6944266. PMID 25570634